CLINICAL TRIAL: NCT05377853
Title: Advanced Spatiomotor Rehabilitation for Navigation in Blindness & Visual Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smith-Kettlewell Eye Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EY024056
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Blindness; Blindness, Acquired; Low Vision; Blindness, Complete
Keywords: blindness; plasticity; spatial memory; training; navigation
MeSH Terms: conditions — Blindness; Vision, Low

STUDY DESIGN:
Intervention Model Description: Multiple regression analyses with life history and vision-related clinical factors as covariates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blindness history (Experimental): Since this is a regression analysis, all participants are assigned to the same Arm with blindness history and the demographics as covariates.
  Interventions: Behavioral: Cognitive-Kinesthetic Navigational Training

INTERVENTIONS:
Behavioral: Cognitive-Kinesthetic Navigational Training — Training with tactile maps to improve spatial memory capability for enhanced navigational capabilities.

SUMMARY:
One of the most challenging tasks for blind and visually impaired individuals is navigation through a complex environment. The goal of the present multidisciplinary study is to increase spatial-cognition abilities in people who are blind or visually impaired through training with the previously-developed Cognitive-Kinesthetic Rehabilitation Training to improve navigation, and to investigate the resultant neuroplastic brain reorganization through multimodal brain imaging.

In accordance with National Eye Institute (NEI) strategic goals, this multidisciplinary project will promote the development of well-informed new approaches to navigational rehabilitation, memory enhancement and cross-modal brain plasticity to benefit 'cutting edge' fields of mobile assistive technologies, vision restoration and memory facilitation for the aging brain.

DETAILED DESCRIPTION:
The investigators propose a radical new multidisciplinary approach to navigation training in blindness and visual impairment. Successful navigation requires the development of an accurate and flexible mental, or cognitive, map of the navigational space and of the route trajectory required to travel from the current to the target location. The Cognitive-Kinesthetic (C-K) Rehabilitation Training that the PI has developed in the preceding period utilizes a unique form of blind memory-guided drawing to develop cognitive mapping to a high level of proficiency. Particular reliance must be placed on such mental maps (supported only by tactile and auditory inputs), and on the ability to use them effectively for spatiomotor control, when vision with its built-in spatial functionality is lost. There is, however, a fundamental gap in the practice of Orientation and Mobility (O&M), which is the lack of a specific emphasis on enhancement of these cognitive roots of spatiomotor activity, despite their known importance for navigation in the visually impaired.

The investigators therefore propose a rigorous multidisciplinary approach to this issue, which lies at the intersection of the fields of spatiomotor rehabilitation, blindness assessment technologies, and brain function, each a focus of one Specific Aim. To train the spatial cognition abilities underlying successful navigation, the current proposal aims to translate the power of the C-K Rehabilitation Training to the domain of navigation. The blind and visually impaired trainees will quickly learn how to generate precise and stable cognitive maps of haptically explored raised-line images or tactile maps, and how to use the formed cognitive maps to confidently guide both drawing 'hand navigation' on a map-scale, and whole-body blind navigation on the macro-scale. Once translated to navigation, the preliminary data show that this efficient and enjoyable training will rapidly and sustainably enhance spatial cognition functions both for improved navigation performance and for enhancement of more general spatial cognitive skills. Beyond its practical advantages, the rapid and effective training protocol will also serve as an efficient tool to drive and study training-based neuroplasticity mechanisms through a comprehensive whole-brain multimodal brain imaging platform.

ELIGIBILITY:
Inclusion Criteria:

Behavioral Studies:

* Vision from < 20/500 to NLP (No Light Perception)

Brain Imaging Studies:

* Vision from < 20/500 to NLP
* Within average gender range for height +/-1 standard deviation
* Within average gender range for weight +/-1 standard deviation
* Comfortable with MRI procedures

Exclusion Criteria:

Behavioral Studies:

* Neurological deficits
* Inability to normally control lower or upper extremities
* Inability to hear and understand instructions.

Brain Imaging Studies:

* All standard MRI exclusion criteria, such as having any metallic objects in the body, or being too large to fit or operate comfortably in the scanner bore.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in blind map drawing speed from pre-training (Pre) to immediate post-training (Post1) timepoints | 6-10 days
  The trajectory of the drawing hand while performing memory-guided navigational tasks will be electronically recorded for assessment of from Pre to Post1 change in terms of drawing speed in cm/s.
  Note: The three timepoints of the study are:
  * Pre: Immediately before the 5-day Cognitive-Kinesthetic training period
  * Post1: Immediately after the 5-day Cognitive-Kinesthetic training period
  * Post2: Within 3-6 months after Post1, without any training intervening between Post1 and Post2
  The time frames for changes and maintenance assessment are given as ranges to allow for scheduling logistics but represent a single interval per participant for each measure.
Maintenance of change in blind map drawing speed from Post1 to extended post-training (Post2) timepoints | 3-6 months
  The trajectory of the drawing hand while performing memory-guided navigational tasks will be assessed for Post1 to Post2 change in drawing speed in cm/s.
Change in blind map drawing errors from Pre to Post1 timepoints | 6-10 days
  The trajectory of the drawing hand while performing memory-guided navigational tasks will be assessed for Pre to Post1 change in navigation drawing errors in terms of number of incorrect turns.
Maintenance of change in blind map drawing errors from Post1 to Post2 timepoints | 3-6 months
  The trajectory of the drawing hand while performing memory-guided navigational tasks will be assessed for Post1 to Post2 change in navigation drawing errors in terms of number of incorrect turns.
Change in total navigation time during blind macro-scale navigation of the shortest path from Pre to Post1 timepoints | 6-10 days
  A tactile map of the virtual layout will be explored and memorized; then, using the formed memory representation of the map, the participants will mentally plan the shortest route between two verbally-provided points on a street map, and walk along that route in the iPhone-encoded Virtual Environment within an Empty Real Space (iVEERS) system developed for this proposal. The iVEERS recorded shortest-path navigation trajectories will be assessed for Pre to Post1 change in total navigation time in s.
Maintenance of change in number of total navigation time during blind navigation of the shortest path at macro-scale from Post1 to Post2 timepoints | 3-6 months
  A tactile map of the virtual layout will be explored and memorized; then, using the formed memory representation of the map, the participants will mentally plan the shortest route between two verbally-provided points on a street map, and walk along that route in the iPhone-encoded Virtual Environment within an Empty Real Space (iVEERS) system developed for this proposal. The iVEERS recorded shortest-path navigation trajectories will be assessed for Post1 to Post2 change in terms of total navigation time measured in s.
Change in total number of contact errors during blind macro-scale navigation from Pre to Post1 timepoints | 6-10 days
  A tactile map of the virtual layout will be explored and memorized; then, using the formed memory representation of the map, the participants will mentally plan the shortest route between two verbally-provided points on a street map, and walk along that route in the iPhone-encoded Virtual Environment within an Empty Real Space (iVEERS) system developed for this proposal. The iVEERS recorded shortest-path navigation trajectories will be assessed for Pre to Post1 change in terms of total number of contact errors.
Maintenance of change in total number of contact errors during blind macro-scale navigation from Post1 to Post2 timepoints | 3-6 months
  A tactile map of the virtual layout will be explored and memorized; then, using the formed memory representation of the map, the participants will mentally plan the shortest route between two verbally-provided points on a street map, and walk along that route in the iPhone-encoded Virtual Environment within an Empty Real Space (iVEERS) system developed for this proposal. The iVEERS recorded shortest-path navigation trajectories will be assessed for Post1 to Post2 change in number of contact errors.
Change in functional MRI (fMRI) activation in the cortical navigation network | 6-10 days
  Whole-brain fMRI will be run to measure activation in the cortical navigation network while the participant plans the shortest paths between two locations based on their memory representations of explored raised-line tactile maps. The change in average activation in the cortical navigation network will be assessed from the Pre to Post1 timepoints in z-score units.
Maintenance of change in fMRI activation in the cortical navigation network | 3-6 months
  Whole-brain fMRI will be run to measure activation in the cortical navigation network while the participant plans the shortest paths between two locations based on their memory representations of explored raised-line tactile maps. The maintenance in average activation in the cortical navigation network will be assessed from the Post1 to Post2 timepoints in z-score units.
Change in functional MRI (fMRI) activation in the spatial working memory network | 6-10 days
  Whole-brain fMRI will be run to measure activation in the spatial working memory network while the participant plans the shortest paths between two locations based on their memory representations of explored raised-line tactile maps. The change in average activation in the spatial working memory network will be assessed from the Pre to Post1 timepoints in z-score units.
Maintenance of change in fMRI activation in the spatial working memory network | 3-6 months
  Whole-brain fMRI will be run to measure activation in the spatial working memory network while the participant plans the shortest paths between two locations based on their memory representations of explored raised-line tactile maps. The change in average activation in the spatial working memory network will be assessed from the Post1 to Post2 timepoints in z-score units.
Change in Granger causal connectivity (GCC) density in the cortical navigation network | 6-10 days
  The changes of the GC connectivity density in the navigation network from the Pre to Post1 will be assessed in terms of the connectivity density index, defined as the ratio of the number of significant GC connections to the number of network nodes.
Maintenance of change in GCC density in the cortical navigation network | 3-6 months
  The changes of the GC connectivity density in the navigation network from the Post1 to Post2 will be assessed in terms of the connectivity density index, defined as the ratio of the number of significant GC connections to the number of network nodes.

SECONDARY OUTCOMES:
Transfer of training to untrained spatio-cognitive abilities | 6-10 days
  The transfer of the training effect to untrained spatio-cognitive abilities will be assessed for a Pre to Post1 change in terms of the score on the Cognitive Test for the Blind (CTB) of the McCarron-Dial Comprehensive Vocational Evaluation System in its standardized IQ-style units.
Maintenance of transfer of training to untrained spatio-cognitive abilities | 3-6 months
  The maintenance of the training effect to untrained spatio-cognitive abilities will be assessed for a Post1 to Post2 change on the Cognitive Test for the Blind (CTB) of the McCarron-Dial Comprehensive Vocational Evaluation System measured in its standardized IQ-style units.
Change in Diffusion Tensor Imaging (DTI) in the cortical navigation network | 6-10 days
  DTI will be used to assess the change in average voxelwise Fractional Anisotropy (FA) throughout the pathways of the cortical navigation network from the Pre to Post1 timepoints in FA z-score units.
Maintenance of change in Diffusion Tensor Imaging (DTI) in the cortical navigation network | 3-6 months
  DTI will be used to assess the change in average voxelwise FA throughout the pathways of the cortical navigation network from the Post1 to Post2 timepoints in FA z-score units.
Change in mobility self-assessment | 3-6 months
  The Kuyk Mobility Function Questionnaire for blindness and profound visual impairment will be used to assess the change in effects of training on everyday mobility from the Pre to the Post2 timepoints in terms of its standardized score.

OTHER OUTCOMES:
Age | Pre-training timepoint
  The covariate of age of the participants will be measured in years.
Gender | Pre-training timepoint.
  The covariate of gender of the participants will be measured in three categorical values (male, intermediate, female).
Current level of vision | Pre-training timepoint
  The covariate of current level of vision of the participants will be measured with the Bailey-Lovey eyechart in Snellen units.
Age of onset of current level of vision | Pre-training timepoint
  The covariate of age of onset of the current level of vision across of the participant will be measured in years.
Duration of full vision | Pre-training timepoint
  The covariate of duration of full vision of the participants will be measured in years.
Duration of Orientation and Mobility (O&M) training | Pre-training timepoint
  The covariate of O&M training of the participants will be measured in years.

CONTACTS AND LOCATIONS:
Overall Officials: Lora T Likova, Principal Investigator — Senior Scientist
Locations (1):
- Smith-Kettlewell Eye Research Institute, San Francisco, California, United States

REFERENCES:
- [Result] Likova LT, Cacciamani L. Transfer of Learning in People Who Are Blind: Enhancement of Spatial-Cognitive Abilities Through Drawing. J Vis Impair Blind. 2018 Jul 1;112(4):385-397. doi: 10.1177/0145482x1811200405. PMID 33223582
- [Result] Likova LT, Mineff KN, Nicholas SC. Mental Visualization in the Cerebellum: Rapid Non-motor Learning at Sub-Lobular and Causal Network Levels. Front Syst Neurosci. 2021 Sep 10;15:655514. doi: 10.3389/fnsys.2021.655514. eCollection 2021. PMID 34566588
- [Result] Likova LT. A Cross-Modal Perspective on the Relationships between Imagery and Working Memory. Front Psychol. 2013 Jan 18;3:561. doi: 10.3389/fpsyg.2012.00561. eCollection 2012. PMID 23346061
- [Result] Likova LT, Tyler CW, Cacciamani L, Mineff K, Nicholas S. The Cortical Network for Braille Writing in the Blind. IS&T Int Symp Electron Imaging. 2016;2016:10.2352/ISSN.2470-1173.2016.16.HVEI-095. doi: 10.2352/ISSN.2470-1173.2016.16.HVEI-095. Epub 2016 Feb 14. PMID 28890944
- [Result] Cacciamani L, Likova LT. Memory-guided drawing training increases Granger causal influences from the perirhinal cortex to V1 in the blind. Neurobiol Learn Mem. 2017 May;141:101-107. doi: 10.1016/j.nlm.2017.03.013. Epub 2017 Mar 24. PMID 28347878
- [Result] Likova LT, Mei M, Mineff KN, Nicholas SC. Learning face perception without vision: Rebound learning effect and hemispheric differences in congenital vs late-onset blindness. IS&T Int Symp Electron Imaging. 2019 Jan 13;2019:2371-23713. doi: 10.2352/ISSN.2470-1173.2019.12.HVEI-237. PMID 31633079
- [Result] Likova LT. Drawing enhances cross-modal memory plasticity in the human brain: a case study in a totally blind adult. Front Hum Neurosci. 2012 May 14;6:44. doi: 10.3389/fnhum.2012.00044. eCollection 2012. PMID 22593738